CLINICAL TRIAL: NCT01958463
Title: Transplantation of Fecal Microbiota for Clostridium Difficile Infection
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TASMC-12-ZH-500-CTIL
Record Dates: First submitted 2013-10-06; First posted 2013-10-09 (Estimated); Last update posted 2013-10-09 (Estimated); Status verified 2013-10

CONDITIONS: Clostridium Difficile Infection
Keywords: Clostridium Difficile Infection; Fecal Microbiota Transplantation
MeSH Terms: conditions — Clostridium Infections | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Fecal microbiota transplantation (Experimental): Fecal microbiota transplantation during colonoscopy.
  Interventions: Procedure: Fecal Microbiota transplantation.

INTERVENTIONS:
Procedure: Fecal Microbiota transplantation. — Fecal Microbiota transplantation during colonoscopy.

SUMMARY:
Recent data have demonstrated beneficial health outcomes of microbiota transplantation for the treatment of Clostridium Difficile infection.

The investigators propose testing whether fecal transplantation from a healthy donor can lead to a recovery from Clostridium Difficile recurrent/treatment-resistant infection.

DETAILED DESCRIPTION:
Infections by Clostridium Difficile are common both in the community and among hospitalized patients. It is mostly prevalent following an antibiotic treatment. In recent years the investigators are witnessing an increase in severity, incidence and treatment-resistant cases.

Treatment-resistant infection or recurrent infection put the patient at risk for severe complications, such as perforation, septic shock, megacolon and even death.

New antibiotic treatments such as Rifaximin and Fidaxomicin are not yet available for routine use in Israel.

It is known that normal intestinal microbiota protect against Clostridium Difficile infections, and as early as 1958, researchers have demonstrated that a transplantation of fecal microbiota had a beneficial effect on Clostridium Difficile Infection.

In fact, previous data show that microbiota transplantation during colonoscopy, in patients with treatment-resistant infection or recurrent infections, is an effective method with a 90% success rate in a single treatment.

The investigators propose testing whether fecal transplantation from a healthy donor can lead to a recovery from Clostridium Difficile infection.

ELIGIBILITY:
Inclusion Criteria:

* age>18 years.
* A negative pregnancy test at inclusion, and a commitment to use contraception for a period of six months from the date of transplant.
* At least one of the following conditions :

  1. An evidence of Clostridium infection recurrence within 6 months after completion of antibiotic course acceptable, which will include at least 10 days of treatment Bmtronidzol a total dose of 500 mg x3 per day and / or Bonkomitzin dose of at least 125 mg 4x a day .

     Recurrence of infection is defined clinical and laboratory :
     * ≥ 3 diarrhea per day for at least two days in a row or ≥ 8 loose stools a day for 48 hours.
     * a positive stool test for Clostridium Difficile toxin, or PCR / antigen detection.
  2. First infection not responding to antibiotics (at least 10 days Metronidazole dosage of 1500 mg per day , or Bonkomitzin total dose of at least 500 mg per day).
  3. A first infection in a patient who is intolerant or allergic to Lonkomitzin and metronidazole.

Exclusion Criteria:

* Participation in another clinical study.
* Inability to provide informed consent.
* A pregnant woman or breastfeeding.
* Severe neutropenia - below 500 neutrophils (blood counts).
* A significant immunosuppression (SCID, CVID, GVHD, using different preparations Aimonosofrsibiim , including prolonged corticosteroid therapy at doses equivalent to ≥ 20 mg prednisone per day for more than 4 weeks).
* Status of SIRS or hemodynamic/respiratory instability.
* Toxic Megacolon, ischemic colitis, Fulminant colitis or a higher than usual risk of colon perforatin during colonoscopy.
* HBV infection or hepatitis C or HIV.
* The use of antibiotics for the treatment of another disease at the time of inclusion.
* A history of previous or current autoimmune disease, a progressive/an uncontrolled disease of the kidney/liver/hematological system/endocrine system/ heart/neurological system, or a metabolic disease.
* An addiction to alcohol or drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2013-11; Primary Completion 2015-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Clinical remission | 8 weeks after treatment
  Less than 3 bowel movements a day

SECONDARY OUTCOMES:
Negative lab test for Clostridium Difficile | 8 weeks after treatment
  No evidence for Clostridium Difficile in stool test.

CONTACTS AND LOCATIONS:
Overall Officials: Zmir Halpern, MD, Principal Investigator — Tel-Aviv Sourasky Medical Center
Locations (1):
- Gastroenterology Institute, Tel Aviv, Israel, Israel